CLINICAL TRIAL: NCT01319175
Title: Hip-Flexion Strength Training: Can Elastic Bands Induce a Relevant Effect?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Allocation: Randomized | Masking: Single
Other Study IDs: H-3-2010-062
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2010-07

CONDITIONS: Hip Flexion Strength
Keywords: hip flexion strength training; elastic bands; external resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Training group (Experimental)
  Interventions: Other: Hip flexion strength training

INTERVENTIONS:
Other: Hip flexion strength training

SUMMARY:
Strength training of the hip flexors using elastic bands can induce an effect on isometric hip strength of at least 15 %.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (more than 2.5 h/week) individuals

Exclusion Criteria:

* Injury in the lower back or legs within the last 6 months.
* Systematic strength training of the hip flexors more than once a week within the last 6 months before the study was initiated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Isometric hip flexion strength | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Metropol, Campus Raadmandsmarken, Copenhagen, Denmark